CLINICAL TRIAL: NCT01739348
Title: A Randomized, Placebo Controlled, Parallel-Group, Double Blind Efficacy and Safety Trial of MK-8931 With a Long Term Double-Blind Extension in Subjects With Mild to Moderate Alzheimer's Disease (Protocol No. MK-8931-017-10)(Also Known as SCH 900931, P07738)
Brief Title: An Efficacy and Safety Trial of Verubecestat (MK-8931) in Mild to Moderate Alzheimer's Disease (P07738)
Acronym: EPOCH
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P07738; MK-8931-017 (Other: Merck Protocol Number); 2011-003151-20 (EudraCT Number); 132229 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2012-11-29; First posted 2012-12-03 (Estimated); Results first posted 2018-05-16 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-09

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — verubecestat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm A. Verubecestat 12 mg [Part I]; 12 mg [Part II] (Experimental): [Part I] Verubecestat 12 mg once daily for 78 weeks in Study Part I (Base Study). [Part II] Participants completing Study Part I and continuing to Study Part II (Extension Study) receive Verubecestat 12 mg once daily for an additional 260 weeks.
  Interventions: Drug: Verubecestat (Part I and Part II)
- Arm B. Verubecestat 40 mg [Part I]; 40 mg [Part II] (Experimental): [Part I] Verubecestat 40 mg once daily for 78 weeks in Study Part I (Base Study). [Part II] Participants completing Study Part I and continuing to Study Part II (Extension Study) receive Verubecestat 40 mg once daily for an additional 260 weeks.
  Interventions: Drug: Verubecestat (Part I and Part II)
- Arm C. Verubecestat 60mg/40mg [Part I]; 40 mg [Part II] (Experimental): [Part I] Verubecestat 60 mg once daily until the first IA in Study Part I (Base Study). Following IA, participants in this group were switched to Verubecestat 40 mg once daily, for the remainder of Study Part I (total dosing period: 78 weeks). [Part II] Participants completing Study Part I and continuing to Study Part II (Extension Study) receive Verubecestat 40 mg once daily for an additional 260 weeks.
  Interventions: Drug: Verubecestat (Part I and Part II)
- Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II] (Placebo Comparator): [Part I] Placebo once daily for 78 weeks in Study Part I (Base Study). [Part II] Participants completing Study Part I and continuing to Study Part II (Extension Study) receive Verubecestat 40 mg once daily for an additional 260 weeks.
  Interventions: Drug: Placebo (Part I); Drug: Verubecestat (Part II)

INTERVENTIONS:
Drug: Verubecestat (Part I and Part II) — Single 12 mg verubecestat tablet once daily, taken orally
  Other Names: SCH 900931
  Arms: Arm A. Verubecestat 12 mg [Part I]; 12 mg [Part II]
Drug: Verubecestat (Part I and Part II) — Single 40 mg verubecestat tablet once daily, taken orally
  Other Names: SCH 900931
  Arms: Arm B. Verubecestat 40 mg [Part I]; 40 mg [Part II]
Drug: Verubecestat (Part I and Part II) — Single 60 or 40 mg verubecestat tablet once daily, taken orally
  Other Names: SCH 900931
  Arms: Arm C. Verubecestat 60mg/40mg [Part I]; 40 mg [Part II]
Drug: Placebo (Part I) — Single placebo tablet matching verubecestat treatment once daily, taken orally
  Arms: Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II]
Drug: Verubecestat (Part II) — Single 40 mg verubecestat tablet once daily, taken orally
  Other Names: SCH 900931
  Arms: Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II]

SUMMARY:
This study consists of two parts, Part I and Part II. The purpose of Part I of the study is to assess the efficacy and safety of verubecestat (MK-8931) compared with placebo administered for 78 weeks in the treatment of Alzheimer's Disease (AD). The primary study hypotheses for Part I are that at least one verubecestat dose is superior to placebo at 78 weeks of treatment with respect to change from baseline in Alzheimer's Disease Assessment Scale Cognitive Subscale (ADAS-Cog) score and that at least one verubecestat dose is superior to placebo at 78 weeks of treatment with respect to change from baseline in Alzheimer's Disease Cooperative Study Activities of Daily Living Inventory (ADCS-ADL) score. The first approximately 400 participants entering Part I of the study are identified as the Safety Cohort. Participants who complete Part I of the study may choose to participate in Part II, which is a long term double-blind extension to assess efficacy and safety of verubecestat administered for up to an additional 260 weeks.

DETAILED DESCRIPTION:
Two substudies are included in Part I of the study: 1) a medical imaging substudy to evaluate changes in brain amyloid protein load using positron emission tomography (PET) and an amyloid tracer ([18F]flutemetamol); and 2) a cerebrospinal fluid (CSF) biomarker substudy to evaluate changes in CSF concentrations of amyloid-β related peptides, total tau, and phosphorylated tau (p-tau). The substudies will be conducted only at designated investigational sites. Participants are not required to take part in a substudy in order to take part in the larger trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable AD based on both a) the National Institute of Neurological and Communicative Diseases and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria and b) the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR) criteria for AD
* AD is of mild to moderate severity
* Clear history of cognitive and functional decline over at least one year that is either a) documented in medical records or b) documented by history from an informant who knows the subject well
* Able to read at a 6th grade level or equivalent, and must have a history of academic achievement and/or employment sufficient to exclude mental retardation
* If a participant is receiving an acetylcholinesterase inhibitor, memantine, medical food/supplement (e.g., vitamin E) and/or herbal medications for AD, the dose must have been stable for at least three months before Screening, and the participant must be willing to remain on the same dose for the duration of the trial. Participants may need to be on AD treatments in accordance with local requirements
* Participant must have a reliable and competent trial partner/caregiver who must have a close relationship with the subject

Inclusion Criteria for Extension Period (Part II):

* Tolerated study drug and completed the initial 78-week period of the trial (Part I)
* Participant must have a reliable and competent trial partner who must have a close relationship with the subject

Exclusion Criteria:

* History of stroke
* Evidence of a neurological disorder other than the disease being studied (i.e., probable AD)
* History of seizures or epilepsy within the last 5 years before Screening
* Evidence of a clinically relevant or unstable psychiatric disorder, excluding major depression in remission
* Participant is at imminent risk of self-harm or of harm to others
* History of alcoholism or drug dependency/abuse within the last 5 years before Screening
* Participant does not have a magnetic resonance imaging (MRI) scan obtained within 12 months of Screening and is unwilling or not eligible to undergo an MRI scan at the Screening Visit. With Sponsor approval, a head computed tomography (CT) scan may be substituted for MRI scan to evaluate eligibility
* History of hepatitis or liver disease that has been active within the six months prior to Screening Visit
* Recent or ongoing, uncontrolled, clinically significant medical condition within 3 months of the Screening Visit (e.g., diabetes, hypertension, thyroid or endocrine disease, congestive heart failure, angina, cardiac or gastrointestinal disease, dialysis, or abnormal renal function) other than the condition being studied such that participation in the trial would pose a significant medical risk to the subject. Controlled co-morbid conditions are not exclusionary if stable within three months of the Screening Visit
* History or current evidence of long QT syndrome, corrected QT (QTc) interval ≥470 milliseconds (for male subjects) or ≥480 milliseconds (for female subjects), or torsades de pointes
* History of malignancy occurring within the five years before Screening, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or localized prostate carcinoma; or malignancy which has been treated with potentially curative therapy with no evidence of recurrence for ≥3 year post-therapy
* Clinically significant vitamin B12 or folate deficiency in the six months before Screening Visit
* Use of any investigational drugs within 30 days (or longer depending on drug) before Screening or participation in studies involving repeated cognitive testing within 30 days before Screening. Participation in an observational study, such as those involving annual cognitive assessments and/or neuroimaging, may be allowed if approved by Sponsor
* History of a hypersensitivity reaction to more than three drugs
* Has tested positive for human immunodeficiency virus (HIV)
* Close family member (including the caregiver, the spouse or any children) who is among the personnel of the investigational or sponsor staff directly involved with this trial

Additional Exclusion Criteria for Safety Cohort:

* History of an ongoing medical condition that has been poorly controlled within 6 months of the Screening Visit (e.g., hypotension, diabetes, hypertension, cerebrovascular disease, thyroid disease, endocrine disturbance, congestive heart failure, cardiac or gastrointestinal disease, dialysis, or abnormal renal function) other than the condition being studied such that a subject's participation in the trial would pose a significant medical risk
* History of congestive heart failure (moderate or greater severity), myocardial infarction, heart surgery, syncope, bradycardia, or clinically significant hypotension within one year before Screening

Exclusion Criteria for Extension Period (Part II):

* Participant is at imminent risk of self-harm or of harm to others
* Has developed a recent or ongoing, uncontrolled, clinically significant medical condition other than AD
* Has history of or has developed during Part I evidence of long QT syndrome, QTc interval ≥470 milliseconds (for male subjects) or ≥480 milliseconds (for female subjects), or torsades de pointes
* Has developed a form of dementia that is not AD

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2211 (Actual)
Dates: Start 2012-11-30 (Actual); Primary Completion 2017-04-14 (Actual); Study Completion 2017-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Sur C, Adamczuk K, Scott D, Kost J, Sampat M, Buckley C, Farrar G, Newton B, Suhy J, Bennacef I, Egan MF. Evaluation of 18F-flutemetamol amyloid PET image analysis parameters on the effect of verubecestat on brain amlyoid load in Alzheimer's disease. Mol Imaging Biol. 2022 Dec;24(6):862-873. doi: 10.1007/s11307-022-01735-z. Epub 2022 Jul 7. PMID 35794343
- [Derived] Dockendorf MF, Jaworowicz D, Humphrey R, Anderson M, Breidinger S, Ma L, Taylor T, Dupre N, Jones C, Furtek C, Kantesaria B, Bateman KP, Woolf E, Egan MF, Stone JA. A Model-Based Approach to Bridging Plasma and Dried Blood Spot Concentration Data for Phase 3 Verubecestat Trials. AAPS J. 2022 Apr 6;24(3):53. doi: 10.1208/s12248-022-00682-5. PMID 35384522
- [Derived] Sur C, Kost J, Scott D, Adamczuk K, Fox NC, Cummings JL, Tariot PN, Aisen PS, Vellas B, Voss T, Mahoney E, Mukai Y, Kennedy ME, Lines C, Michelson D, Egan MF. BACE inhibition causes rapid, regional, and non-progressive volume reduction in Alzheimer's disease brain. Brain. 2020 Dec 1;143(12):3816-3826. doi: 10.1093/brain/awaa332. PMID 33253354
- [Derived] Sergott RC, Raji A, Kost J, Sur C, Jackson S, Locco A, Patel A, Furtek C, Mattson B, Egan MF. Retinal Optical Coherence Tomography Metrics Are Unchanged in Verubecestat Alzheimer's Disease Clinical Trial but Correlate with Baseline Regional Brain Atrophy. J Alzheimers Dis. 2021;79(1):275-287. doi: 10.3233/JAD-200735. PMID 33252075
- [Derived] Egan MF, Mukai Y, Voss T, Kost J, Stone J, Furtek C, Mahoney E, Cummings JL, Tariot PN, Aisen PS, Vellas B, Lines C, Michelson D. Further analyses of the safety of verubecestat in the phase 3 EPOCH trial of mild-to-moderate Alzheimer's disease. Alzheimers Res Ther. 2019 Aug 7;11(1):68. doi: 10.1186/s13195-019-0520-1. PMID 31387606
- [Derived] Egan MF, Kost J, Tariot PN, Aisen PS, Cummings JL, Vellas B, Sur C, Mukai Y, Voss T, Furtek C, Mahoney E, Harper Mozley L, Vandenberghe R, Mo Y, Michelson D. Randomized Trial of Verubecestat for Mild-to-Moderate Alzheimer's Disease. N Engl J Med. 2018 May 3;378(18):1691-1703. doi: 10.1056/NEJMoa1706441. PMID 29719179
- [Derived] Kennedy ME, Stamford AW, Chen X, Cox K, Cumming JN, Dockendorf MF, Egan M, Ereshefsky L, Hodgson RA, Hyde LA, Jhee S, Kleijn HJ, Kuvelkar R, Li W, Mattson BA, Mei H, Palcza J, Scott JD, Tanen M, Troyer MD, Tseng JL, Stone JA, Parker EM, Forman MS. The BACE1 inhibitor verubecestat (MK-8931) reduces CNS beta-amyloid in animal models and in Alzheimer's disease patients. Sci Transl Med. 2016 Nov 2;8(363):363ra150. doi: 10.1126/scitranslmed.aad9704. PMID 27807285

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part I began by enrolling approximately 50 participants per arm (200 total). Enrollment continued until the first 200 participants reached 13 weeks treatment; total enrollment at that time: ~400. For these ~400 participants (Safety Cohort), an interim analysis (IA) was conducted to assess safety. Following IA, enrollment continued (Main Cohort).
Pre-assignment Details: 2211 participants were randomized in Part I, with 2210 receiving treatment. As planned per protocol, no participants were randomized to the Verubecestat 60 mg arm (Arm C) in the Main Cohort. Participants completing Part I were eligible to continue to Part II. The trial was terminated early and did not complete as planned.
Period: Part I (Base Study)
Arm/Group | Arm A. Verubecestat 12 mg [Part I]; 12 mg [Part II] | Arm B. Verubecestat 40 mg [Part I]; 40 mg [Part II] | Arm C. Verubecestat 60mg/40mg [Part I]; 40 mg [Part II] | Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II]
Started | 703 | 700 | 103 | 705
Treated | 702 | 700 | 103 | 705
Completed | 501 | 497 | 77 | 516
Not Completed | 202 | 203 | 26 | 189
Not completed — Adverse Event | 41 | 52 | 8 | 33
Not completed — Death | 10 | 7 | 2 | 8
Not completed — Lack of Efficacy | 3 | 8 | 0 | 7
Not completed — Lost to Follow-up | 4 | 2 | 4 | 4
Not completed — Non-Compliance with Study Drug | 3 | 2 | 0 | 0
Not completed — Physician Decision | 10 | 7 | 1 | 4
Not completed — Protocol Violation | 2 | 0 | 1 | 2
Not completed — Screen Failure | 2 | 0 | 0 | 0
Not completed — Site Discontinued Study Participation | 1 | 3 | 0 | 0
Not completed — Study Terminated by Sponsor | 72 | 73 | 0 | 86
Not completed — Participant Moved | 4 | 3 | 1 | 7
Not completed — Trial Partner/Caregiver Withdrew Consent | 27 | 25 | 2 | 18
Not completed — Withdrawal by Subject | 23 | 21 | 7 | 20
Period: Part II (Extension Study)
Arm/Group | Arm A. Verubecestat 12 mg [Part I]; 12 mg [Part II] | Arm B. Verubecestat 40 mg [Part I]; 40 mg [Part II] | Arm C. Verubecestat 60mg/40mg [Part I]; 40 mg [Part II] | Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II]
Started | 379 (Number started refers only to participants completing Part I, volunteering to continue to Part II.) | 366 (Number started refers only to participants completing Part I, volunteering to continue to Part II.) | 61 (Number started refers only to participants completing Part I, volunteering to continue to Part II.) | 396 (Number started refers only to participants completing Part I, volunteering to continue to Part II.)
Treated | 379 | 365 | 61 | 394
Completed | 0 | 0 | 0 | 0
Not Completed | 379 | 366 | 61 | 396
Not completed — Adverse Event | 10 | 11 | 7 | 26
Not completed — Death | 3 | 3 | 2 | 6
Not completed — Lack of Efficacy | 1 | 5 | 0 | 1
Not completed — Lost to Follow-up | 3 | 4 | 0 | 1
Not completed — Non-Compliance with Study Drug | 0 | 0 | 0 | 1
Not completed — Physician Decision | 7 | 11 | 6 | 12
Not completed — Study Terminated by Sponsor | 329 | 315 | 34 | 323
Not completed — Participant Moved | 3 | 3 | 0 | 3
Not completed — Trial Partner/Caregiver Withdrew Consent | 18 | 12 | 8 | 16
Not completed — Withdrawal by Subject | 5 | 2 | 4 | 7

BASELINE CHARACTERISTICS:
Population: All randomized participants in Study Part I (Base Study)
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A. Verubecestat 12 mg [Part I]; 12 mg [Part II] | Arm B. Verubecestat 40 mg [Part I]; 40 mg [Part II] | Arm C. Verubecestat 60mg/40mg [Part I]; 40 mg [Part II] | Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II] | Total
Number analyzed (Participants) | 703 | 700 | 103 | 705 | 2211
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.2 (7.4) | 71.8 (7.6) | 72.3 (7.4) | 72.4 (7.6) | 71.8 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 383 | 403 | 56 | 376 | 1218
  Male | 320 | 297 | 47 | 329 | 993
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 0 | 3 | 7
  Asian | 118 | 125 | 11 | 115 | 369
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 13 | 2 | 7 | 30
  White | 566 | 547 | 88 | 578 | 1779
  More than one race | 4 | 4 | 2 | 0 | 10
  Unknown or Not Reported | 6 | 8 | 0 | 2 | 16
Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) Score [Mean (Standard Deviation); unit: Score on a Scale] — ADAS-Cog measures cognition by assessing 11 metrics impaired in Alzheimer's Disease (AD): speech; speech comprehension; word finding; word recall; object/finger naming; orientation; obeying commands; ideational praxis; constructional praxis; word recognition; and remembering instruction. For each metric, scores range from 0 (no impairment) to (depending on the metric) either 5 (8 metrics), 8, 10, or 12 (1 metric each); higher scores indicate more severe impairment. Individual scores sum to a total ADAS-Cog score, ranging from 0-70. Higher total scores indicate greater cognitive impairment. Population: All randomized participants (Part I) with a baseline and ≥1 within-analysis-window ADAS-Cog observation subsequent to ≥1 dose of study drug (Full Analysis Set [FAS] population).
  Score on a Scale
    number analyzed (Participants) | 681 | 672 | 97 | 694 | 2144
    (all) | 21.4 (7.5) | 21.3 (7.6) | 20.6 (6.2) | 21.7 (7.6) | 21.42 (7.49)
Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL) Score [Mean (Standard Deviation); unit: Score on a Scale] — The ADCS-ADL score measures the performance of activities of daily living, calculated from a 24-question survey. For each of the 24 questions, scores range from 0 (no independence) to (depending on the question) either 2 (1 question), 3 (17 questions), 4 (5 questions), or 5 (1 question), with higher scores indicating greater independence in activity performance. Scores from individual questions are summed into a total ADCS-ADL score, with total scores ranging from 0 to 78. Lower scores indicate less independence in activity performance. Population: All randomized participants (Part I) with a baseline and ≥1 within-analysis-window observation for ADCS-ADL subsequent to ≥1 dose of study drug (FAS population).
  Score on a Scale
    number analyzed (Participants) | 677 | 668 | 98 | 686 | 2129
    (all) | 63.0 (9.5) | 62.9 (9.8) | 63.5 (10.3) | 62.1 (10.4) | 62.74 (9.93)
Clinical Dementia Rating Sum of Boxes (CDR-SB) Score [Mean (Standard Deviation); unit: Score on a Scale] — The CDR-SB score is a clinical rating of global cognitive function, comprised of 6 domains including: memory; orientation; judgment and problem solving; community affairs; home and hobbies; and personal care. For each domain, the degree of impairment is assessed by a semi-structured interview of the participant as well as the participant's caregiver. For each domain, potential scores range from 0 (no impairment) to 3 (severe impairment). Individual domain scores sum to the total CDR-SB score, with total scores ranging from 0-18. Higher scores indicate more severe cognitive impairment. Population: All randomized participants (Part I) with a baseline and ≥1 within-analysis-window observation for CDR-SB subsequent to ≥1 dose of study drug (FAS population).
  Score on a Scale
    number analyzed (Participants) | 660 | 643 | 91 | 673 | 2067
    (all) | 5.4 (2.1) | 5.3 (2.1) | 5.5 (2.3) | 5.6 (2.3) | 5.43 (2.17)
Total Hippocampal Volume [Mean (Standard Deviation); unit: Microliters] — Total Hippocampal Volume (THV) was measured by volumetric magnetic resonance imaging (vMRI). Population: All randomized participants (Part I) with a baseline and ≥1 within-analysis-window observation for THV subsequent to ≥1 dose of study drug (FAS population).
  Microliters
    number analyzed (Participants) | 332 | 307 | 55 | 346 | 1040
    (all) | 5894.1 (1231.5) | 5823.4 (1189.9) | 5653.5 (1148.4) | 5800.7 (1069.2) | 5829.4 (1162.6)
Cerebrospinal Fluid (CSF) Total Tau Concentration [Mean (Standard Deviation); unit: picograms (pg)/mL] — Total Tau concentration in the cerebrospinal fluid (CSF) was monitored as a measure of brain tau pathology. Population: All randomized participants (Part I) with a baseline and ≥1 within-analysis-window observation for CSF Total Tau subsequent to ≥1 dose of study drug (FAS population). Per protocol, CSF Total Tau concentration was analyzed as part of a substudy in Part I, with testing occurring at select trial sites.
  picograms (pg)/mL
    number analyzed (Participants) | 38 | 57 | 12 | 41 | 148
    (all) | 206.7 (90.4) | 231.5 (113.9) | 268.6 (136.2) | 246.2 (192.9) | 232.2 (137.3)
[18F]Flutemetamol Positron Emission Tomography (PET) Standard Uptake Value Ratio (SUVR) [Mean (Standard Deviation); unit: SUVR] — [18F]Flutemetamol PET SUVR measures brain cortical amyloid load. The PET tracer [18F]Flutemetamol was given intravenously (IV). After 90 minutes, participants receive 4 PET scans. Using the PET scan images, regional SUVRs are calculated for brain regions of interest (ROIs), defined as the ratio of pixel intensities at a specific ROI compared to a reference region (RR; subcortical white matter). Regional SUVRs are averaged to compute a composite SUVR. Higher composite SUVR values indicate increased amyloid load. Population: All randomized participants with a baseline and ≥1 within-analysis-window SUVR observation subsequent to ≥1 dose of study drug (FAS population). SUVR testing occurred at select sites as a Part I substudy. Per protocol, SUVR was not analyzed for the 200 participants enrolled before IA (all arms) and all participants receiving 60mg Verubecestat.
  SUVR
    number analyzed (Participants) | 20 | 10 | 0 | 14 | 44
    (all) | 0.89 (0.10) | 0.87 (0.11) |  | 0.88 (0.11) | 0.88 (0.10)
Neuropsychiatric Inventory (NPI) Score [Mean (Standard Deviation); unit: Score on a Scale] — NPI is a clinical assessment of psychiatric status, covering 12 domains. Based on an interview of the participant's caregiver, each domain is assessed for symptom frequency [range: 1 (occasional) to 4 (very frequent)] and severity [range: 1 (mild) to 3 (severe)]. Domain scores [range: 0 to 12] are calculated as the product of the frequency and severity scores (i.e. frequency x severity); if no symptoms are present, domain score is 0. The 12 domain scores sum to a total NPI score [range: 0 (no symptoms in any domain) to 144]. Higher scores reflect more severe psychiatric impairment. Population: All randomized participants (Part I) with a baseline and ≥1 within-analysis-window NPI observation subsequent to ≥1 dose of study drug (FAS population).
  Score on a Scale
    number analyzed (Participants) | 682 | 679 | 100 | 691 | 2152
    (all) | 8.7 (10.5) | 8.2 (9.8) | 6.9 (9.5) | 9.2 (11.6) | 8.64 (10.6)
Mini-Mental State Examination (MMSE) Score [Mean (Standard Deviation); unit: Score on a Scale] — The MMSE is a cognitive assessment of 5 domains including: orientation; attention; memory; language; and constructional praxis. These domains are assessed with 11 total questions related to the participant. Participants are scored based on the number of correct responses; depending on the question, potential scores range from 0 (no correct response) to either 1 (4 questions), 2 (1 question), 3 (3 questions), or 5 (3 questions). Scores from each question are summed to the total MMSE score, with total scores ranging from 0-30. Higher scores indicate better cognitive performance. Population: All randomized participants (Part I) with a baseline and ≥1within-analysis-window MMSE observation subsequent to ≥1 dose of study drug (FAS population).
  Score on a Scale
    number analyzed (Participants) | 660 | 648 | 98 | 679 | 2085
    (all) | 20.4 (3.3) | 20.2 (3.3) | 20.6 (3.3) | 20.3 (3.2) | 20.3 (3.3)

OUTCOME MEASURES:

1. Primary Outcome: [Part I (Base Study)] Change From Baseline in the Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) Score
Description: Least squares mean change from baseline at week 78 was assessed for the ADAS-Cog score. ADAS-Cog measures cognition by assessing 11 metrics impaired in Alzheimer's Disease (AD): speech; speech comprehension; word finding; word recall; object/finger naming; orientation; obeying commands; ideational praxis; constructional praxis; word recognition; and remembering instruction. For each metric, scores range from 0 (no impairment) to (depending on the metric) either 5 (8 metrics), 8, 10, or 12 (1 metric each); higher scores indicate more severe impairment. Individual scores sum to a total ADAS-Cog score, ranging from 0-70. Higher total scores indicate greater cognitive impairment and AD severity. Further, increases in AD severity over time would be reflected by increases in ADAS-Cog score.
Time Frame: Baseline and week 78
Population: All randomized participants with a baseline and ≥1 within-analysis-window ADAS-Cog observation subsequent to ≥1 dose of study drug (FAS population). Per protocol, the 200 participants enrolled before IA (all arms) and all participants receiving 60mg Verubecestat (Arm C) were excluded.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Arm A. Verubecestat 12 mg [Part I]; 12 mg [Part II] | Arm B. Verubecestat 40 mg [Part I]; 40 mg [Part II] | Arm C. Verubecestat 60mg/40mg [Part I]; 40 mg [Part II] | Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II]
Number analyzed (Participants) | 631 | 626 | 0 | 644
Score on a Scale | 7.9 [7.2 to 8.6] | 8.0 [7.3 to 8.7] |  | 7.7 [7.0 to 8.4]
Statistical Analysis 1: Comparison: Arm A. Verubecestat 12 mg [Part I]; 12 mg [Part II] vs Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II]; Test type: Superiority; p = 0.6287, Longitudinal ANCOVA; Difference in Least Squares Mean = 0.2, 97.51% CI 2-sided [-0.9 to 1.3]
Statistical Analysis 2: Comparison: Arm B. Verubecestat 40 mg [Part I]; 40 mg [Part II] vs Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II]; Test type: Superiority; p = 0.4625, Longitudinal ANCOVA; Difference in Least Squares Mean = 0.4, 97.51% CI 2-sided [-0.8 to 1.5]

2. Primary Outcome: [Part I (Base Study)] Change From Baseline in Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL) Score
Description: Least squares mean change from baseline at week 78 was assessed for the ADCS-ADL score. The ADCS-ADL score measures the performance of activities of daily living, calculated from a 24-question survey. For each of the 24 questions, scores range from 0 (no independence) to (depending on the question) either 2 (1 question), 3 (17 questions), 4 (5 questions), or 5 (1 question), with higher scores indicating greater independence in activity performance. Scores from individual questions are summed into a total ADCS-ADL score, with total scores ranging from 0 to 78. Lower scores indicate less independence in activity performance and, as a result, greater AD severity. Further, increases in AD severity over time would be reflected by decreases in ADCS-ADL score.
Time Frame: Baseline and week 78
Population: All randomized participants with a baseline and ≥1 within-analysis-window ADCS-ADL observation subsequent to ≥1 dose of study drug (FAS population). Per protocol, the 200 participants enrolled before IA (all arms) and all participants receiving 60mg Verubecestat (Arm C) were excluded.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Arm A. Verubecestat 12 mg [Part I]; 12 mg [Part II] | Arm B. Verubecestat 40 mg [Part I]; 40 mg [Part II] | Arm C. Verubecestat 60mg/40mg [Part I]; 40 mg [Part II] | Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II]
Number analyzed (Participants) | 627 | 622 | 0 | 636
Score on a Scale | -8.4 [-9.5 to -7.4] | -8.2 [-9.2 to -7.1] |  | -8.9 [-9.9 to -8.0]
Statistical Analysis 1: Comparison: Arm A. Verubecestat 12 mg [Part I]; 12 mg [Part II] vs Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II]; Test type: Superiority; p = 0.4925, Longitudinal ANCOVA; Difference in Least Squares Means = 0.5, 97.51% CI 2-sided [-1.1 to 2.1]
Statistical Analysis 2: Comparison: Arm B. Verubecestat 40 mg [Part I]; 40 mg [Part II] vs Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II]; Test type: Superiority; p = 0.3221, Longitudinal ANCOVA; Difference in Least Squares Means = 0.7, 97.51% CI 2-sided [-0.9 to 2.3]

3. Primary Outcome: [Part II (Extension Study)] Change From Baseline in Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) Score
Description: Mean change from baseline at week 104 was assessed for the ADAS-Cog score. ADAS-Cog measures cognition by assessing 11 metrics impaired in Alzheimer's Disease (AD): speech; speech comprehension; word finding; word recall; object/finger naming; orientation; obeying commands; ideational praxis; constructional praxis; word recognition; and remembering instruction. For each metric, scores range from 0 (no impairment) to (depending on the metric) either 5 (8 metrics), 8, 10, or 12 (1 metric each); higher scores indicate more severe impairment. Individual scores sum to a total ADAS-Cog score, ranging from 0-70. Higher total scores indicate greater cognitive impairment and AD severity. Further, increases in AD severity over time would be reflected by increases in ADAS-Cog score. Per study protocol, the baseline measurement to be used was the baseline measurement obtained in Part I.
Time Frame: Baseline and week 104
Population: All randomized participants continuing to Part II, with a baseline and ≥1 within-analysis-window ADAS-Cog observation subsequent to ≥1 dose of study drug (FAS population), having an ADAS-Cog observation at week 104. Per protocol, the 200 participants enrolled before IA (all arms) and all participants receiving 60mg Verubecestat were excluded.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Arm A. Verubecestat 12 mg [Part I]; 12 mg [Part II] | Arm B. Verubecestat 40 mg [Part I]; 40 mg [Part II] | Arm C. Verubecestat 60mg/40mg [Part I]; 40 mg [Part II] | Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II]
Number analyzed (Participants) | 207 | 208 | 0 | 216
Score on a Scale | 10.1 (9.9) | 8.5 (9.5) |  | 9.6 (9.5)

4. Primary Outcome: [Part II (Extension Study)] Change From Baseline in Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL) Score
Description: Mean change from baseline at week 104 was assessed for the ADCS-ADL score. The ADCS-ADL score measures the performance of activities of daily living, calculated from a 24-question survey. For each of the 24 questions, scores range from 0 (no independence) to (depending on the question) either 2 (1 question), 3 (17 questions), 4 (5 questions), or 5 (1 question), with higher scores indicating greater independence in activity performance. Scores from individual questions are summed into a total ADCS-ADL score, with total scores ranging from 0 to 78. Lower scores indicate less independence in activity performance and, as a result, greater AD severity. Further, increases in AD severity over time would be reflected by decreases in ADCS-ADL score. Per study protocol, the baseline measurement to be used was the baseline measurement obtained in Part I.
Time Frame: Baseline and week 104
Population: All randomized participants continuing to Part II, with a baseline and ≥1 within-analysis-window ADCS-ADL observation subsequent to ≥1 dose of study drug (FAS population), having an ADCS-ADL observation at week 104. Per protocol, the 200 participants enrolled before IA (all arms) and all participants receiving 60mg Verubecestat were excluded.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Arm A. Verubecestat 12 mg [Part I]; 12 mg [Part II] | Arm B. Verubecestat 40 mg [Part I]; 40 mg [Part II] | Arm C. Verubecestat 60mg/40mg [Part I]; 40 mg [Part II] | Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II]
Number analyzed (Participants) | 207 | 209 | 0 | 216
Score on a Scale | -10.7 (13.7) | -9.2 (12.7) |  | -9.3 (12.0)

5. Primary Outcome: [Part I (Base Study)] Number of Participants Who Experienced an Adverse Event
Description: The number of participants experiencing an adverse event (AE) in Part I was assessed. An AE is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to this medicinal product. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product is also an AE.
Time Frame: Up to week 80 (up to 2 weeks following cessation of study treatment in Part I)
Population: Includes all randomized participants in Part I receiving ≥1 dose of trial treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A. Verubecestat 12 mg [Part I]; 12 mg [Part II] | Arm B. Verubecestat 40 mg [Part I]; 40 mg [Part II] | Arm C. Verubecestat 60mg/40mg [Part I]; 40 mg [Part II] | Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II]
Number analyzed (Participants) | 702 | 700 | 103 | 705
Participants | 630 | 646 | 90 | 579

6. Primary Outcome: [Part II (Extension Study)] Number of Participants Who Experienced an Adverse Event
Description: The number of participants experiencing an adverse event (AE) in Part II was assessed. An AE is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to this medicinal product. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product is also an AE.
Time Frame: From week 78 (end of treatment in Part I) up to week 262 of Part II
Population: Includes all randomized participants continuing to Part II, receiving ≥1 dose of trial treatment in Part II. For included participants, the data reflect AEs occurring in Part II only.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A. Verubecestat 12 mg [Part I]; 12 mg [Part II] | Arm B. Verubecestat 40 mg [Part I]; 40 mg [Part II] | Arm C. Verubecestat 60mg/40mg [Part I]; 40 mg [Part II] | Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II]
Number analyzed (Participants) | 379 | 365 | 61 | 394
Participants | 240 | 230 | 51 | 264

7. Primary Outcome: [Part I (Base Study)] Number of Participants Who Discontinued From Study Drug Due to an Adverse Event
Description: The number of participants discontinuing from study drug due to an AE in Part I was assessed. An AE is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to this medicinal product. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product is also an AE.
Time Frame: Up to week 78
Population: Includes all randomized participants in Part I receiving ≥1 dose of trial treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A. Verubecestat 12 mg [Part I]; 12 mg [Part II] | Arm B. Verubecestat 40 mg [Part I]; 40 mg [Part II] | Arm C. Verubecestat 60mg/40mg [Part I]; 40 mg [Part II] | Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II]
Number analyzed (Participants) | 702 | 700 | 103 | 705
Participants | 57 | 64 | 12 | 42

8. Primary Outcome: [Part II (Extension Study)] Number of Participants Who Discontinued From Study Drug Due to an Adverse Event
Description: The number of participants discontinuing from study drug due to an AE in Part II was assessed. An AE is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to this medicinal product. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product is also an AE.
Time Frame: From week 78 (end of treatment in Part I) up to week 260 of Part II
Population: Includes all randomized participants continuing to Part II, receiving ≥1 dose of trial treatment in Part II. For included participants, the data reflect treatment discontinuations occurring in Part II only.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A. Verubecestat 12 mg [Part I]; 12 mg [Part II] | Arm B. Verubecestat 40 mg [Part I]; 40 mg [Part II] | Arm C. Verubecestat 60mg/40mg [Part I]; 40 mg [Part II] | Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II]
Number analyzed (Participants) | 379 | 365 | 61 | 394
Participants | 10 | 9 | 6 | 29

9. Secondary Outcome: [Part I (Base Study)] Change From Baseline in Clinical Dementia Rating Sum of Boxes (CDR-SB) Score
Description: Least squares mean change from baseline at week 78 was assessed for CDR-SB score. The CDR-SB score is a clinical rating of global cognitive function, comprised of 6 domains including: memory; orientation; judgment and problem solving; community affairs; home and hobbies; and personal care. For each domain, the degree of impairment is assessed by a semi-structured interview of the participant as well as the participant's caregiver. For each domain, potential scores range from 0 (no impairment) to 3 (severe impairment). Scores from each individual domain are summed to the total CDR-SB score, with total scores ranging from 0-18. Higher scores indicate more severe cognitive impairment. Further, increases in cognitive impairment would be reflected by increases in CDR-SB score.
Time Frame: Baseline and week 78
Population: All randomized participants with a baseline and ≥1 within-analysis-window CDR-SB observation subsequent to ≥1 dose of study drug (FAS population). Per protocol, the 200 participants enrolled before IA (all arms) and all participants receiving 60mg Verubecestat (Arm C) were excluded.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Arm A. Verubecestat 12 mg [Part I]; 12 mg [Part II] | Arm B. Verubecestat 40 mg [Part I]; 40 mg [Part II] | Arm C. Verubecestat 60mg/40mg [Part I]; 40 mg [Part II] | Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II]
Number analyzed (Participants) | 611 | 600 | 0 | 623
Score on a Scale | 2.1 [1.8 to 2.3] | 2.1 [1.9 to 2.4] |  | 2.1 [1.9 to 2.3]
Statistical Analysis 1: Comparison: Arm A. Verubecestat 12 mg [Part I]; 12 mg [Part II] vs Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II]; Test type: Superiority; p = 0.8426, Longitudinal ANCOVA; Difference in Least Squares Means = 0.0, 97.51% CI 2-sided [-0.4 to 0.3]
Statistical Analysis 2: Comparison: Arm B. Verubecestat 40 mg [Part I]; 40 mg [Part II] vs Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II]; Test type: Superiority; p = 0.8264, Longitudinal ANCOVA; Difference in Least Squares Means = 0.0, 97.51% CI 2-sided [-0.3 to 0.4]

10. Secondary Outcome: [Part I (Base Study)] Percent Change From Baseline in Total Hippocampal Volume (THV)
Description: Least squares mean percent change from baseline at week 78 was calculated for Total Hippocampal Volume (THV) as measured by volumetric magnetic resonance imaging (vMRI). Longitudinal analysis of within-participant THV is computed using a change analysis algorithm using tensor-based morphometry. This technique produces one measure of volume change calculated from the registration of serial vMRI scans at the follow-up time point relative to baseline. Negative percent changes from baseline indicate decreases in THV (i.e. increased hippocampal atrophy).
Time Frame: Baseline and week 78
Population: All randomized participants with a baseline and ≥1 within-analysis-window THV observation subsequent to ≥1 dose of study drug (FAS population). Per protocol, the 200 participants enrolled prior to IA (all arms) and all participants receiving 60mg Verubecestat (Arm C) were excluded.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Arm A. Verubecestat 12 mg [Part I]; 12 mg [Part II] | Arm B. Verubecestat 40 mg [Part I]; 40 mg [Part II] | Arm C. Verubecestat 60mg/40mg [Part I]; 40 mg [Part II] | Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II]
Number analyzed (Participants) | 308 | 281 | 0 | 308
Percent Change | -5.6 [-5.9 to -5.4] | -5.7 [-5.9 to -5.4] |  | -5.0 [-5.2 to -4.7]
Statistical Analysis 1: Comparison: Arm A. Verubecestat 12 mg [Part I]; 12 mg [Part II] vs Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II]; Test type: Superiority; p = 0.0005, Longitudinal ANCOVA; Difference in Least Squares Means = -0.6, 97.51% CI 2-sided [-1.0 to -0.2]
Statistical Analysis 2: Comparison: Arm B. Verubecestat 40 mg [Part I]; 40 mg [Part II] vs Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II]; Test type: Superiority; p = 0.0002, Longitudinal ANCOVA; Difference in Least Squares Means = -0.7, 97.51% CI 2-sided [-1.1 to -0.3]

11. Secondary Outcome: [Part I (Base Study)] Fold Change From Baseline in Cerebrospinal Fluid (CSF) Total Tau
Description: Least squares mean fold change from baseline at week 78 was calculated for Total Tau concentration in CSF, a measure of brain tau pathology. Per protocol, CSF Total Tau concentration was analyzed as part of a substudy in Part I, with testing occurring only at select trial sites. Least squares mean fold change from baseline >1 indicates increased Total Tau concentration in the CSF.
Time Frame: Baseline and week 78
Population: All randomized participants with a baseline and ≥1 within-analysis-window CSF Total Tau observation subsequent to ≥1 dose of study drug (FAS population). Per protocol, the 200 participants enrolled prior to IA (all arms) and all participants receiving 60mg Verubecestat (Arm C) were excluded.
Measure: Least Squares Mean (95% Confidence Interval); unit: Fold Change
Arm/Group | Arm A. Verubecestat 12 mg [Part I]; 12 mg [Part II] | Arm B. Verubecestat 40 mg [Part I]; 40 mg [Part II] | Arm C. Verubecestat 60mg/40mg [Part I]; 40 mg [Part II] | Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II]
Number analyzed (Participants) | 32 | 46 | 0 | 33
Fold Change | 1.02 [0.96 to 1.08] | 1.04 [0.99 to 1.09] |  | 1.07 [1.01 to 1.13]
Statistical Analysis 1: Comparison: Arm A. Verubecestat 12 mg [Part I]; 12 mg [Part II] vs Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II]; Test type: Superiority; p = 0.2138, Longitudinal ANCOVA; Ratio of Fold Change from Baseline = 0.95, 95% CI 2-sided [0.87 to 1.04]
Statistical Analysis 2: Comparison: Arm B. Verubecestat 40 mg [Part I]; 40 mg [Part II] vs Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II]; Test type: Superiority; p = 0.4330, Longitudinal ANCOVA; Ratio of Fold Change from Baseline = 0.97, 95% CI 2-sided [0.90 to 1.05]

12. Secondary Outcome: [Part I (Base Study)] Change From Baseline in Cortical Amyloid Load Assessed by [18F]Flutemetamol PET Standard Uptake Value Ratio (SUVR)
Description: Least squares mean change from baseline at week 78 was calculated for SUVR, a measure of brain cortical amyloid load. Per protocol, SUVR was analyzed as part of a substudy in Part I, with testing occurring only at select trial sites. Participants receive the PET tracer [18F]Flutemetamol (IV). After 90 minutes, participants receive 4 PET scans (5 minutes each in duration). Using these PET scan images, specific brain ROIs (frontal, temporal, and parietal lobes; anterior and posterior cingulate and precuneus) are used to calculate regional SUVRs, defined as the relative ratio of pixel intensities at a specific ROI compared to a reference region (RR; subcortical white matter). These regional SUVRs are then averaged to compute a composite cortical SUVR for each participant. Higher composite cortical SUVR values indicate increased amyloid load, with negative changes in composite cortical SUVR over time indicating decreases in brain amyloid load.
Time Frame: Baseline and week 78
Population: All randomized participants with a baseline and ≥1 within-analysis-window SUVR observation subsequent to ≥1 dose of study drug (FAS population). Per protocol, the 200 participants enrolled prior to IA (all arms) and all participants receiving 60mg Verubecestat did not receive SUVR testing and were excluded.
Measure: Least Squares Mean (95% Confidence Interval); unit: SUVR
Arm/Group | Arm A. Verubecestat 12 mg [Part I]; 12 mg [Part II] | Arm B. Verubecestat 40 mg [Part I]; 40 mg [Part II] | Arm C. Verubecestat 60mg/40mg [Part I]; 40 mg [Part II] | Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II]
Number analyzed (Participants) | 20 | 10 | 0 | 14
SUVR | -0.02 [-0.04 to -0.01] | -0.04 [-0.06 to -0.03] |  | 0.00 [-0.01 to 0.01]
Statistical Analysis 1: Comparison: Arm A. Verubecestat 12 mg [Part I]; 12 mg [Part II] vs Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II]; Test type: Superiority; p = 0.0066, Longitudinal ANCOVA; Difference in Least Squares Means = -0.03, 95% CI 2-sided [-0.05 to 0.00]
Statistical Analysis 2: Comparison: Arm B. Verubecestat 40 mg [Part I]; 40 mg [Part II] vs Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II]; Test type: Superiority; p < 0.0001, Longitudinal ANCOVA; Difference in Least Squares Means = -0.04, 95% CI 2-sided [-0.06 to -0.02]

13. Secondary Outcome: [Part I (Base Study)] Percentage of Participants Achieving Responder Status
Description: The percentage of participants achieving responder status at week 78 was assessed. To determine which participants were considered responders, a linear regression was conducted at the participant level, yielding an estimated 78-week rate of change (i.e., a slope) for each participant with respect to ADAS-Cog and ADCS-ADL. To be declared a responder, a participant must have: 1) ADAS-Cog and ADCS-ADL observations at baseline and 78 weeks of treatment; 2) an ADAS-Cog slope > 4.0 over 78 weeks, and 3) an ADCS-ADL slope > -6.3 over 78 weeks. A participant failing to meet any of these criteria was designated as a non-responder at Week 78.
Time Frame: Week 78
Population: All randomized participants in Part I receiving ≥1 dose of trial treatment. Per protocol, the first 200 participants enrolled prior to IA (across all arms) and all participants receiving 60mg Verubecestat (Arm C) were excluded from analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm A. Verubecestat 12 mg [Part I]; 12 mg [Part II] | Arm B. Verubecestat 40 mg [Part I]; 40 mg [Part II] | Arm C. Verubecestat 60mg/40mg [Part I]; 40 mg [Part II] | Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II]
Number analyzed (Participants) | 652 | 652 | 0 | 653
Percentage of Participants | 20.1 | 19.6 |  | 19.3

14. Secondary Outcome: [Part I (Base Study)] Change From Baseline in Neuropsychiatric Inventory (NPI) Score
Description: Least squares mean change from baseline at week 78 was assessed for NPI score. NPI is a clinical assessment of psychiatric status, covering 12 domains: delusion; hallucination; agitation/aggression; depression/dysphoria; anxiety; elation/euphoria; apathy/indifference; disinhibition; irritability/lability; aberrant motor behavior; sleep/nighttime behaviors; and appetite/eating disorders. Based on an interview of the participant's caregiver, each domain is assessed for symptom frequency [range: 1 (occasional) to 4 (very frequent)] and severity [range: 1 (mild) to 3 (severe)]. Domain scores [range: 0 to 12] are calculated as the product of the frequency and severity scores (i.e. frequency x severity); if no symptoms are present, domain score is 0. The 12 domain scores sum to a total NPI score [range: 0 (no symptoms in any domain) to 144]. Higher scores reflect more severe psychiatric impairment, with increases in impairment reflected by increases in NPI score.
Time Frame: Baseline and week 78
Population: All randomized participants with a baseline and ≥1 within-analysis-window NPI observation subsequent to ≥1 dose of study drug (FAS population). Per protocol, the 200 participants enrolled prior to IA (all arms) and all participants receiving 60mg Verubecestat (Arm C) were excluded.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Arm A. Verubecestat 12 mg [Part I]; 12 mg [Part II] | Arm B. Verubecestat 40 mg [Part I]; 40 mg [Part II] | Arm C. Verubecestat 60mg/40mg [Part I]; 40 mg [Part II] | Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II]
Number analyzed (Participants) | 632 | 631 | 0 | 639
Score on a Scale | 3.4 [2.5 to 4.4] | 3.8 [2.8 to 4.8] |  | 2.7 [1.7 to 3.7]
Statistical Analysis 1: Comparison: Arm A. Verubecestat 12 mg [Part I]; 12 mg [Part II] vs Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II]; Test type: Superiority; p = 0.2949, Longitudinal ANCOVA; Difference in Least Squares Means = 0.7, 95% CI 2-sided [-0.6 to 2.1]
Statistical Analysis 2: Comparison: Arm B. Verubecestat 40 mg [Part I]; 40 mg [Part II] vs Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II]; Test type: Superiority; p = 0.1372, Longitudinal ANCOVA; Difference in Least Squares Means = 1.1, 95% CI 2-sided [-0.4 to 2.6]

15. Secondary Outcome: [Part I (Base Study)] Change From Baseline in Mini-Mental State Examination (MMSE) Score
Description: Least squares mean change from baseline at week 78 was assessed for MMSE score. The MMSE is a cognitive assessment of 5 domains including: orientation; attention; memory; language; and constructional praxis. These domains are assessed over the course of 11 total questions related to the participant. Participants are scored based on the number of correct responses; depending on the question, potential scores range from 0 (no correct response) to either 1 (4 questions), 2 (1 question), 3 (3 questions), or 5 (3 questions). Scores from each question are summed to the total MMSE score, with total scores ranging from 0-30. Higher scores indicate better cognitive performance. Further, deterioration in cognitive performance would be reflected by decreases in MMSE score.
Time Frame: Baseline and week 78
Population: All randomized participants with a baseline and ≥1 within-analysis-window MMSE observation subsequent to ≥1 dose of study drug (FAS population). Per protocol, the 200 participants enrolled prior to IA (all arms) and all participants receiving 60mg Verubecestat (Arm C) were excluded.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Arm A. Verubecestat 12 mg [Part I]; 12 mg [Part II] | Arm B. Verubecestat 40 mg [Part I]; 40 mg [Part II] | Arm C. Verubecestat 60mg/40mg [Part I]; 40 mg [Part II] | Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II]
Number analyzed (Participants) | 610 | 600 | 0 | 628
Score on a Scale | -3.9 [-4.3 to -3.6] | -3.6 [-4.0 to -3.3] |  | -4.1 [-4.5 to -3.8]
Statistical Analysis 1: Comparison: Arm A. Verubecestat 12 mg [Part I]; 12 mg [Part II] vs Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II]; Test type: Superiority; p = 0.4721, Longitudinal ANCOVA; Difference in Least Squares Means = 0.2, 95% CI 2-sided [-0.3 to 0.7]
Statistical Analysis 2: Comparison: Arm B. Verubecestat 40 mg [Part I]; 40 mg [Part II] vs Arm D. Placebo [Part I]; Verubecestat 40 mg [Part II]; Test type: Superiority; p = 0.0599, Longitudinal ANCOVA; Difference in Least Squares Means = 0.5, 95% CI 2-sided [0.0 to 1.0]

ADVERSE EVENTS:
Time Frame: [Part I]: Up to week 80 of Part I (up to 2 weeks following cessation of study treatment in Part I); [Part II]: From week 78 (end of treatment in Part I) up to week 262 of Study Part II
Description: [Part I] Includes all randomized participants in Study Part I (Base Study) receiving ≥1 dose of trial treatment. [Part II] Includes all randomized participants continuing to Study Part II (Extension Study) receiving ≥1 dose of trial treatment in Part II. For Part II-specific arms, only the AEs occurring during study Part II are reported.
Groups:
- Arm A. Verubecestat 12 mg [Part I]: [Part I] Verubecestat 12 mg once daily for 78 weeks in Study Part I (Base Study).
- Arm B. Verubecestat 40 mg [Part I]: [Part I] Verubecestat 40 mg once daily for 78 weeks in Study Part I (Base Study).
- Arm C. Verubecestat 60mg/40mg [Part I]: [Part I] Verubecestat 60 mg once daily until the first IA in Study Part I (Base Study). Following IA, participants in this group were switched to Verubecestat 40 mg once daily, for the remainder of Study Part I (total dosing period: 78 weeks).
- Arm D. Placebo [Part I]: [Part I] Placebo once daily for 78 weeks in Study Part I (Base Study).
- Arm A. Verubecestat 12 mg [Part II]: [Part II] Participants completing Study Part I and continuing to Study Part II (Extension Study) receive Verubecestat 12 mg once daily for an additional 260 weeks.
- Arm B. Verubecestat 40 mg [Part II]; Arm C. Verubecestat 40 mg [Part II]; Arm D. Verubecestat 40 mg [Part II]: [Part II] Participants completing Study Part I and continuing to Study Part II (Extension Study) receive Verubecestat 40 mg once daily for an additional 260 weeks.
Arm/Group | Arm A. Verubecestat 12 mg [Part I] | Arm B. Verubecestat 40 mg [Part I] | Arm C. Verubecestat 60mg/40mg [Part I] | Arm D. Placebo [Part I] | Arm A. Verubecestat 12 mg [Part II] | Arm B. Verubecestat 40 mg [Part II] | Arm C. Verubecestat 40 mg [Part II] | Arm D. Verubecestat 40 mg [Part II]
All-Cause Mortality (participants affected / at risk) | 9/702 | 13/700 | 3/103 | 6/705 | 6/379 | 4/365 | 4/61 | 8/394
Serious Adverse Events (participants affected / at risk) | 134/702 | 162/700 | 24/103 | 121/705 | 57/379 | 56/365 | 22/61 | 69/394
Other Adverse Events (participants affected / at risk) | 408/702 | 440/700 | 66/103 | 337/705 | 135/379 | 102/365 | 37/61 | 144/394
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A. Verubecestat 12 mg [Part I] (N=702) | Arm B. Verubecestat 40 mg [Part I] (N=700) | Arm C. Verubecestat 60mg/40mg [Part I] (N=103) | Arm D. Placebo [Part I] (N=705) | Arm A. Verubecestat 12 mg [Part II] (N=379) | Arm B. Verubecestat 40 mg [Part II] (N=365) | Arm C. Verubecestat 40 mg [Part II] (N=61) | Arm D. Verubecestat 40 mg [Part II] (N=394)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Torsade de pointes (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid cyst (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Corneal oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macular oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trichiasis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulum oesophageal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conduction disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drowning (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Euthanasia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incarcerated hernia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mass (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic cyst (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder empyema (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningoencephalitis herpetic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurosyphilis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 6 (6) | 3 (3) | 5 (5) | 3 (3) | 5 (5) | 3 (3) | 4 (4)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retroperitoneal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tuberculous pleurisy (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fracture displacement (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 5 (5) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prescribed overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ammonia increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood glucose decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose fluctuation (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart rate irregular (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipoprotein (a) increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatic specific antigen increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemic syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Starvation (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atypical fibroxanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (11) | 9 (14) | 1 (1) | 15 (17) | 2 (3) | 3 (3) | 1 (1) | 2 (3)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder transitional cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Borderline mucinous tumour of ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Extradural neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sarcoma uterus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 3 (4) | 2 (2) | 3 (3) | 5 (5) | 1 (1) | 2 (2) | 0 (0)
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 2 (2) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 6 (6) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dementia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 5 (5)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diplegia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 3 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lumbosacral radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Psychomotor skills impaired (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 7 (7) | 13 (15) | 0 (0) | 5 (5) | 1 (1) | 3 (4) | 2 (2) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Abnormal behaviour (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Agitation (Psychiatric disorders) | 4 (5) | 4 (4) | 1 (1) | 0 (0) | 5 (6) | 0 (0) | 1 (2) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Delusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Delusional disorder, persecutory type (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Delusional disorder, unspecified type (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Emotional distress (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Neuropsychiatric symptoms (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Paranoia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psychogenic movement disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal behaviour (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urethral disorder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Noninfective bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal pouch (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A. Verubecestat 12 mg [Part I] (N=702) | Arm B. Verubecestat 40 mg [Part I] (N=700) | Arm C. Verubecestat 60mg/40mg [Part I] (N=103) | Arm D. Placebo [Part I] (N=705) | Arm A. Verubecestat 12 mg [Part II] (N=379) | Arm B. Verubecestat 40 mg [Part II] (N=365) | Arm C. Verubecestat 40 mg [Part II] (N=61) | Arm D. Verubecestat 40 mg [Part II] (N=394)
Anaemia (Blood and lymphatic system disorders) | 8 (8) | 11 (11) | 1 (1) | 6 (6) | 5 (5) | 1 (1) | 4 (5) | 5 (5)
Constipation (Gastrointestinal disorders) | 30 (32) | 27 (29) | 9 (9) | 20 (20) | 13 (14) | 3 (3) | 4 (5) | 10 (10)
Diarrhoea (Gastrointestinal disorders) | 56 (65) | 60 (70) | 4 (9) | 42 (45) | 8 (9) | 8 (8) | 4 (5) | 9 (10)
Bronchitis (Infections and infestations) | 24 (28) | 10 (11) | 6 (7) | 19 (19) | 9 (12) | 5 (5) | 2 (2) | 4 (5)
Urinary tract infection (Infections and infestations) | 61 (79) | 71 (93) | 15 (18) | 56 (68) | 20 (25) | 18 (21) | 5 (6) | 28 (34)
Viral upper respiratory tract infection (Infections and infestations) | 60 (81) | 50 (60) | 5 (5) | 42 (49) | 21 (27) | 11 (12) | 2 (2) | 10 (11)
Contusion (Injury, poisoning and procedural complications) | 25 (31) | 30 (33) | 7 (9) | 21 (27) | 14 (21) | 8 (8) | 2 (2) | 5 (5)
Fall (Injury, poisoning and procedural complications) | 56 (84) | 59 (75) | 8 (8) | 39 (51) | 31 (37) | 19 (25) | 7 (14) | 22 (27)
Weight decreased (Investigations) | 47 (48) | 44 (44) | 7 (7) | 21 (22) | 10 (10) | 8 (8) | 2 (2) | 13 (13)
Decreased appetite (Metabolism and nutrition disorders) | 19 (20) | 30 (31) | 6 (7) | 16 (16) | 4 (4) | 0 (0) | 1 (1) | 10 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 36 (41) | 26 (26) | 4 (5) | 21 (23) | 8 (11) | 7 (8) | 5 (5) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 36 (39) | 46 (49) | 6 (6) | 30 (34) | 8 (8) | 7 (7) | 2 (3) | 6 (6)
Dizziness (Nervous system disorders) | 33 (34) | 56 (70) | 12 (15) | 32 (35) | 9 (9) | 3 (3) | 1 (1) | 8 (10)
Headache (Nervous system disorders) | 42 (48) | 52 (59) | 5 (7) | 41 (58) | 4 (6) | 5 (5) | 2 (2) | 6 (9)
Abnormal dreams (Psychiatric disorders) | 11 (11) | 15 (16) | 6 (6) | 6 (6) | 1 (2) | 1 (1) | 0 (0) | 3 (3)
Agitation (Psychiatric disorders) | 31 (32) | 16 (17) | 5 (7) | 19 (20) | 8 (8) | 5 (5) | 5 (6) | 10 (11)
Anxiety (Psychiatric disorders) | 40 (41) | 47 (51) | 8 (10) | 27 (29) | 6 (6) | 6 (6) | 6 (6) | 8 (8)
Depression (Psychiatric disorders) | 47 (52) | 46 (48) | 9 (9) | 38 (38) | 5 (5) | 6 (6) | 5 (5) | 8 (9)
Insomnia (Psychiatric disorders) | 41 (42) | 33 (33) | 6 (6) | 21 (23) | 12 (12) | 8 (8) | 2 (2) | 10 (10)
Suicidal ideation (Psychiatric disorders) | 39 (42) | 45 (55) | 4 (4) | 24 (26) | 12 (14) | 9 (9) | 2 (2) | 12 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 32 (38) | 26 (27) | 6 (6) | 22 (23) | 7 (9) | 9 (10) | 1 (1) | 13 (14)
Rash (Skin and subcutaneous tissue disorders) | 33 (38) | 26 (31) | 6 (6) | 25 (31) | 7 (7) | 3 (3) | 1 (1) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the sponsor, 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial. The sponsor shall have the right to review and comment with respect to publications, abstracts, slides, and manuscripts and the right to review and comment on the data analysis and presentation.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-01): https://cdn.clinicaltrials.gov/large-docs/48/NCT01739348/Prot_SAP_000.pdf